CLINICAL TRIAL: NCT06400108
Title: Dementia Moves: Protocol for a Pilot Feasibility Study Testing a Physical Rehabilitation Program for Long-Term Care Residents With Moderate to Severe Dementia
Brief Title: Dementia Moves: Protocol for a Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Alzheimer Society of Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-17
Record Dates: First submitted 2024-04-23; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Moderate to Severe Dementia

STUDY DESIGN:
Intervention Model Description: pre-post pilot feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia Moves (Experimental): Dementia Moves is a multi-component exercise intervention that was developed to provide evidence informed exercise-based physical rehabilitation for LTC residents with dementia. The intervention is based on a recent systematic review that examined the effectiveness of physical rehabilitation interventions for LTC residents with dementia and a qualitative study that describes the goals of rehabilitation as described by residents, family members, and staff. The systematic review identified common interventions and their effectiveness, outcome measures, and gaps in the literature, while the qualitative study provided perspective on common goals to determine a future primary outcome of interest.
  Dementia Moves will be delivered to a group of residents (e.g., 4 residents) for 30 minutes, 3 times per week, for a duration of 6 months by a physiotherapist, physiotherapy assistant, and volunteers.
  Interventions: Other: Dementia Moves

INTERVENTIONS:
Other: Dementia Moves — Dementia Moves: Dementia Moves is a multicomponent exercise program that can be individually tailored to the abilities of LTC residents with more advanced dementia and focuses on moderate- to high-intensity strength and balance activities with an aim to improve ADLs. Individualized strategies are implemented throughout the intervention to support and promote participation of individuals with more advanced dementia.
  Each exercise will be individually prescribed for each participant by the physiotherapists (PT) at the beginning of the program. The intensity of the exercise will be adjusted throughout the program by the PT to ensure the target intensity of moderate to high intensity balance and strength exercises. The intervention will be provided face to face in groups of 4 residents with the PT, PTA, and three volunteers. Though the intervention is delivered in a group setting, the specific exercises that the participants complete are individualized based on their abilities.

SUMMARY:
Most long-term care (LTC) residents live with frailty and dementia and the proportion with more advanced cognitive impairment is increasing. Residents with dementia often have limited functional ability to complete their activities of daily living (ADLs) and are vulnerable to further functional decline. Multicomponent exercise can help prevent functional decline, but residents with dementia are less likely to receive it and have not often been included in previous intervention studies. The Dementia Moves intervention was designed to fill this gap. It is an individually tailored multicomponent group exercise program with an aerobic warm-up and a focus on moderate to high intensity functional balance and strength training. This pilot feasibility study will examine the feasibility of delivering Dementia Moves with 16 LTC residents across 2 homes in Nova Scotia (primary outcomes: recruitment, retention, adherence, acceptability, barriers/facilitators to delivery, fidelity; secondary outcomes: ADLs, adverse events). The next step will be to conduct a larger trial to determine the effect of the intervention on ADLs.

Through a parallel cluster randomized controlled trial, investigators will measure the effect of the Dementia Moves program on ADLs and adverse events (i.e., falls, fractures, hospitalizations, emergency department visits) for LTC residents with moderate to severe dementia (i.e., Mini-Mental State Exam of 20 or less).

DETAILED DESCRIPTION:
Background: Most long-term care (LTC) residents live with dementia and the proportion with more advanced cognitive impairment is increasing. Residents with dementia often have limited functional ability to complete their activities of daily living (ADLs) and are vulnerable to further functional decline. Multicomponent exercise can help prevent functional decline, but residents with dementia are less likely to receive it and have not often been included in previous intervention studies. The Dementia Moves intervention was designed to fill this gap. It is an individually tailored multicomponent group exercise program with an aerobic warm-up and a focus on moderate to high intensity functional balance and strength training. Investigators will measure the feasibility and effect of the Dementia Moves program on ADLs for LTC residents with moderate to severe dementia (Mini-Mental State Exam of 20 or less). Investigators hypothesize the intervention will be feasible without modification if 16 individuals are recruited over 6 months, 65% of our sample is retained at 6-months, and 75% of the completed exercises are performed at a moderate to high intensity.

Methods: A pre-post pilot study will be used to assess feasibility, safety (rates of falls and adverse events), and change in ADLs at three- and six-months among LTC residents with moderate to severe dementia. A physiotherapist, physiotherapy assistant, and three volunteers will deliver the group-based exercise program to groups of four residents, three times per week, for six months. Assessments will be completed at three- and six-months. Feasibility outcomes include 1) recruitment over six-months; 2) retention at three- and six-month follow-up; and adherence via 3) attendance and 4) proxy and self-reported ratings of exercise intensity. Investigators will also assess fidelity of the intervention through program audits, and audio diaries and interviews to identify barriers and facilitators to implementation of the intervention.

Discussion: The feasibility of the Dementia Moves intervention will be evaluated in LTC residents with dementia, and investigators will examine rates of falls and adverse events and change in ADLs. Investigators will use the collected information to inform a definitive parallel cluster randomized controlled trial. The feasibility of the Dementia Moves intervention will be evaluated in LTC residents with dementia, and investigators will examine rates of falls and adverse events and change in ADLs. Investigators will use the collected information to inform a definitive parallel cluster randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of any form of dementia as documented in their electronic medical record
2. a Mini-Mental State Exam Score (MMSE) of 20 or less, or Cognitive Performance Scale (CPS) Score of 3 or higher, indicating moderate to severe cognitive impairment.

Exclusion Criteria:

Participants who are receiving end of life care in the LTC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of residents recruited from participating homes | The recruitment will occur over a six-month period,
  Investigators plan to recruit eight residents from each of the two participating homes, distributing our recruitment efforts evenly between them. To manage recruitment efficiently, investigators will alternate our focus between the two homes on a monthly basis. For instance, in the first month, recruitment will be on participants from Home A, then shift our focus to Home B in the second month, and so forth. A target recruitment numbers align with previous studies in long-term care settings for residents with dementia, where successful recruitment has ranged from 12 to 26 residents per home per year. By aiming slightly higher with a total of 16 participants over six months, investigators maintain feasibility while ensuring an adequately sized sample for meaningful analysis.
Participation rates | 3 to 6 months follow-ups.
  Investigators will report the number and percentage of potential participants who are eligible, provide consent, and begin the intervention. The criterion for success is that 80% of eligible participants will complete baseline testing, and attend the first intervention session.
  Number and percentage of participants who complete three- and six-month follow-ups.
  Criteria for success: A total of 13 (81.3%) and 10 (65%) residents will complete three- and six-month follow-ups, respectively.
Attendance rates | 3- and 6-month follow-ups.
  The physiotherapist will take attendance at each exercise session and will document the reason if the resident does not attend (i.e., does not wish to participate, unwell, in hospital, at another activity, or other). Based on the results of previous physical rehabilitation studies for LTC residents with dementia, the criterion for success is the average proportion of exercise sessions attended will be 70%.
Intensity of exercises - resistance and aerobic exercise | 3- and 6-month follow-ups.
  Intensity will be assessed using proxy reports from the study team members and self-reports from the participants. The rate of perceived exertion (RPE) scale used for aerobic and strength exercises which is scored from 0-10, where 0 indicates lower intensity and 10 indicates higher intensity. This information will be recorded by a research assistant throughout the sessions to ensure accurate reporting.
Intensity of exercises - balance | 3- and 6-month follow-ups.
  Intensity will be assessed using proxy reports from the study team members and self-reports from the participants. The Balance Intensity Scale Therapist Reported (BIS-T) and Exerciser Reported (BIS-E) will be used for balance exercises. The BIS-T is scored from 0-100 where a higher number indicates a higher intensity. The BIS-E is scored from 1 to 5 where a higher score indicates more intensity. This information will be recorded by a research assistant throughout the sessions to ensure accurate reporting.

SECONDARY OUTCOMES:
Emergency department visits | three-months prior to baseline, baseline to three-months, and three- to six-month periods.
  The number of visits to the emergency department related and unrelated to the intervention will be reported by the investigators. This includes any visits that may be directly or indirectly related to the intervention, such as those for injuries sustained during exercise sessions or for unrelated health issues. The goal is to provide a comprehensive understanding of the impact of the intervention on residents' health and well-being, including any potential risks or benefits associated with the program.
Activities of daily living (Barthel Index) | baseline at enrollment
  The Barthel Index measures the level of independence in ADLs. The survey consists of 10 performance items (e.g. toilet use, dressing) and each item can be rated on a two, three- or four-point scale indicating the level of help needed for a total of 20 possible points, where a higher score indicates a higher level of functional independence. The survey will be completed by a research assistant through consultation with the nursing staff on each resident's home unit. The Barthel Index is a reliable and valid measure of functional disability and demonstrates excellent inter-rater reliability when used to assess ADLs in LTC homes.
Activities of daily living (interRAI Long-Term Care Facilities Long Form Score) | At enrollment, three- and six-month follow ups
  The interRAI ADL Long Form Scale is a summary scale where each ADL has six possible categories of response ranging from 0 (total independence) to 4 (total dependence) and a score of 8 is assigned if the activity was not performed. The ADL Long Form Scale is the sum of the responses to all seven individual ADL items (bed mobility, transfer, locomotion, dressing, eating, toilet use, personal hygiene) with scores ranging from 0 to 28, where a higher score indicates more dependence. The ADL items that form the scale are collected from the interRAI LTC Facilities Instrument, a valid and reliable comprehensive assessment. It is completed for all LTC residents in Nova Scotia upon admission to the home, every three months thereafter, or if there is a significant change in the resident's health status.
Fall frequency | three-months prior to baseline, baseline to three-months, and three- to six-month periods
  The number of falls that participants experience will be recorded and reported. This information is important for evaluating the effectiveness of the intervention in reducing fall incidents among the study population.
Number of hospitalization | three-months prior to baseline, baseline to three-months, and three- to six-month periods.
  Number of hospitalization will be recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin McArthur, PhD, Principal Investigator — Dalhousie University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lane NE, Wodchis WP, Boyd CM, Stukel TA. Disability in long-term care residents explained by prevalent geriatric syndromes, not long-term care home characteristics: a cross-sectional study. BMC Geriatr. 2017 Feb 10;17(1):49. doi: 10.1186/s12877-017-0444-1. PMID 28183274
- [Background] Helvik AS, Engedal K, Benth JS, Selbaek G. A 52 month follow-up of functional decline in nursing home residents - degree of dementia contributes. BMC Geriatr. 2014 Apr 10;14:45. doi: 10.1186/1471-2318-14-45. PMID 24720782
- [Background] van Doorn C, Gruber-Baldini AL, Zimmerman S, Hebel JR, Port CL, Baumgarten M, Quinn CC, Taler G, May C, Magaziner J; Epidemiology of Dementia in Nursing Homes Research Group. Dementia as a risk factor for falls and fall injuries among nursing home residents. J Am Geriatr Soc. 2003 Sep;51(9):1213-8. doi: 10.1046/j.1532-5415.2003.51404.x. PMID 12919232
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] Ripley S, Alizadehsaravi N, Affoo R, Hunter S, Middleton LE, Moody E, Weeks LE, McArthur C. Resident-, family-, and staff-identified goals for rehabilitation of long-term care residents with dementia: a qualitative study. BMC Geriatr. 2024 Jan 29;24(1):108. doi: 10.1186/s12877-024-04674-2. PMID 38287257
- [Background] Telenius EW, Engedal K, Bergland A. Long-term effects of a 12 weeks high-intensity functional exercise program on physical function and mental health in nursing home residents with dementia: a single blinded randomized controlled trial. BMC Geriatr. 2015 Dec 3;15:158. doi: 10.1186/s12877-015-0151-8. PMID 26630910
- [Background] Slaughter SE, Estabrooks CA, Jones CA, Wagg AS. Mobility of Vulnerable Elders (MOVE): study protocol to evaluate the implementation and outcomes of a mobility intervention in long-term care facilities. BMC Geriatr. 2011 Dec 16;11:84. doi: 10.1186/1471-2318-11-84. PMID 22176583
- [Background] Barisch-Fritz B, Trautwein S, Scharpf A, Krell-Roesch J, Woll A. Effects of a 16-Week Multimodal Exercise Program on Physical Performance in Individuals With Dementia: A Multicenter Randomized Controlled Trial. J Geriatr Phys Ther. 2022 Jan-Mar 01;45(1):3-24. doi: 10.1519/JPT.0000000000000308. PMID 33813533
- [Background] McArthur C, Alizadehsaravi N, Affoo R, Cooke K, Douglas N, Earl M, Flynn T, Ghanouni P, Hunter S, Middleton L, Moody E, Searle S, Smith C, Weeks L. Effectiveness of physical rehabilitation in improving physical functioning and quality of life for long-term-care residents with dementia: a systematic review protocol. JBI Evid Synth. 2023 Jan 1;21(1):207-213. doi: 10.11124/JBIES-22-00096. PMID 36036561
- [Background] Bouwstra H, Smit EB, Wattel EM, van der Wouden JC, Hertogh CMPM, Terluin B, Terwee CB. Measurement Properties of the Barthel Index in Geriatric Rehabilitation. J Am Med Dir Assoc. 2019 Apr;20(4):420-425.e1. doi: 10.1016/j.jamda.2018.09.033. Epub 2018 Nov 16. PMID 30448338
- [Background] Morris JN, Fries BE, Morris SA. Scaling ADLs within the MDS. J Gerontol A Biol Sci Med Sci. 1999 Nov;54(11):M546-53. doi: 10.1093/gerona/54.11.m546. PMID 10619316
- [Background] Glenny C, Stolee P. Comparing the functional independence measure and the interRAI/MDS for use in the functional assessment of older adults: a review of the literature. BMC Geriatr. 2009 Nov 29;9:52. doi: 10.1186/1471-2318-9-52. PMID 19943969
- [Background] Hutchinson AM, Milke DL, Maisey S, Johnson C, Squires JE, Teare G, Estabrooks CA. The Resident Assessment Instrument-Minimum Data Set 2.0 quality indicators: a systematic review. BMC Health Serv Res. 2010 Jun 16;10:166. doi: 10.1186/1472-6963-10-166. PMID 20550719
- [Derived] McArthur C, Alizadehsaravi N, Affoo R, Cooke K, Douglas NF, Earl M, Farlie MK, Flynn T, Ghanouni P, Hunter SW, Grant SM, Middleton LE, Moody E, Smith C, Verlinden L, Weeks LE. Dementia Moves: protocol for a feasibility study testing a physical rehabilitation program for long-term care residents with moderate to severe dementia. Pilot Feasibility Stud. 2025 Jul 26;11(1):104. doi: 10.1186/s40814-025-01685-7. PMID 40713920
- See also: Bennett CA. An evaluation of fall prevention interventions among older adults in a long term care facility. [Internet]. Evaluation of fall prevention interventions among older adults in a long term care facility. University of Southern Mississippi; 201 — http://search.ebscohost.com/login.aspx?direct=true&db=cin20&AN=109794747&site=ehost-live